CLINICAL TRIAL: NCT06013527
Title: Physical Rehabilitation Program for Cardiorespiratory Health and Quality of Life Among Breast Cancer Survivors in UAE - A Randomized Control Trial.
Brief Title: Physical Rehabilitation Program for Cardiorespiratory Health and Quality of Life Among Breast Cancer Survivors in UAE.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Principal Investigator, Fatima Abdul Rashid, Ms., Gulf Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-COHS-STD-95-May-2023
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer survivor; Quality of life; Cardiorespiratory health; Physical rehabilitation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Therapy Intervention (Experimental): The intervention group will receive a structured exercise program which will run for 2 months and a follow-up will be done after 3 months.
  Interventions: Other: Supervised Training; Other: Individually tailored home program
- Control Group (No Intervention): This group will continue with their routine life and will receive standard care given by the hospital.

INTERVENTIONS:
Other: Supervised Training — Two different classes over alternate weeks twice per week :
  1. 60-minute step aerobics class (Given week 1,3,5,7)
  2. 60 minutes circuit training class (Given week 2,4,6,8)
  Each class will include warm-up and cool-down periods both lasting 10-15 min. The exercise period of 30 minutes the maximum target RPE would be set at 14-16 on a 20-point BORG scale, a level of exercise that feels "somewhat hard" or "hard" and coincides with about 86-92% of maximal heart rate, 76-85% of maximal VO 2 and 5-7 metabolic equivalents (METs) ideal for improving the related domains of QoL and Cardiovascular endurance (12). During the first 3 weeks, the participants would exercise at a lower level of RPE (approximately 11-13), to adapt to the training and so that newly recruited participants could also join the group without difficulty.
  Arms: Physical Therapy Intervention
Other: Individually tailored home program — The type of home training would mainly consist of endurance training such as walking, Nordic walking, or aerobic training, but it would also include jumps and leaps like step aerobics to promote bone health. The Participants will be asked to perform these thrice per week.
  Arms: Physical Therapy Intervention

SUMMARY:
This randomized control trial aims to analyze the changes in cardiovascular endurance and quality of life domains for breast cancer survivors in the United Arab Emirates using a long-term 2-month physical rehabilitation program adapted from the BREX protocol.

DETAILED DESCRIPTION:
Cancer is a medical condition where some cells of the body reproduce uncontrollably and metastasize to other parts of the body. The burden of the disease is significantly high both at the global and national levels. In the year 2020, 19.3 million total new cases of cancer were recorded, and cancer deaths were estimated to be 10.0 million, for both males and females. In UAE, cancer was found to be the third leading cause of death. Specifically in UAE, breast cancer was ranked 1 due to its prevalence, incidence, and mortality. Amongst all types of cancers, breast carcinoma is very common among females across the globe which significantly affects their Quality of Life (QoL) with poor cardiovascular tolerance even after the carcinoma has been treated or removed. Thus, the associated morbidity among breast cancer survivors affects all domains of quality of life comprising physical health, psychological health, level of independence, social interactions, and environmental changes.

It is well known that QoL domains are interrelated where physical rehabilitation is of utmost importance as it can help to address all domains. In addition, the "cardiorespiratory systems" are the main functional unit of our circulatory system and provide energy for body movements. Poor cardiovascular endurance has been very commonly reported among breast cancer survivors, which has a direct effect on individuals' level of independence and ability to participate in the social environment thereby adding to overall QoL. Physical rehabilitation forms an important part of breast cancer management pre- and post-surgical. In the pre-surgical phase, rehabilitation can help the individual to sustain the ill effect of post-surgical complications better. However, it is the post-surgical phase that requires more attention and rehabilitation strategies to combat the situation and help the individual regain their functional level near normal. The importance and benefits of physical rehabilitation among breast cancer survivors have been well reported with evidence in the literature.

Integrated structured exercise programs have been defined and prescribed to check their benefits over the QoL domains. In addition, a study reported that while structured exercise programs should focus on improving cardiorespiratory fitness and muscular strength during exercise training, these programs should consider physical activity outside of training, if well-tolerated, to potentially further lower fatigue and improve QOL in cancer survivors. Thus, an individual-centric approach could be more beneficial. Although a recent study reported a higher incidence and prevalence of breast cancer in the UAE population, no published data was found on the application of the recommended exercise regimen, rehabilitation program, and guidelines for breast cancer survivors in the UAE despite a significant level of evidence.

Therefore, the proposed research project aims to improve the QoL domains and Cardiovascular endurance among breast cancer survivors in the United Arab Emirates using physical rehabilitation and recommended exercise programs. An individual-centric approach is intended to maximize the benefits of physical rehabilitation and to match individual needs efficiently.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from breast cancer who have undergone Chemotherapy, Mastectomy, and cleared for post-surgical physical rehabilitation.
* Age group -18 years to 65 years
* Female patients only (gender predisposition)
* Diagnosed with stage I-stage IIIa breast cancer. (As other stages of cancer include metastasis).

Exclusion Criteria:

* Patients diagnosed with prior cardiorespiratory disorders, cognitive dysfunction, and other health problems that would prevent safe participation.
* Active breast cancer patients.
* Participants who engaged in physical activity like the intervention group in any form.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory health | 0-5 months
  A 2-km walk test (UKK walk test, Tampere, Finland) would be done along to evaluate the submaximal Vo2 analysis additionally peak exercise minute ventilation, and direct maximal voluntary ventilation will be assessed to evaluate pulmonary limitation to exercise. This be measured through Spirometry.
Quality of Research | 0-5 months
  The European Organization for Research and Treatment of Cancer (EORTC) questionnaire (EORTC QLQ-C30).

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Abdul Rashid, Principal Investigator — Gulf Medical University
Locations (2):
- United Arab Emirates (2):
  - Thumbay Medical City, Al Jurf, Ajman Emirate
  - Al Tawam, Abu Dhabi

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Rashid FA, Anwar W, Kandakurti PK, Al Qawasmeh KHA, Latif MF, Tirmazy SH, Omara M, Hazari A. Physical rehabilitation program for cardiorespiratory health and quality of life among breast cancer survivors in UAE: a randomized control trial. BMC Cancer. 2025 Apr 16;25(1):705. doi: 10.1186/s12885-025-14005-2. PMID 40241061
- [Derived] Rashid FA, Anwar W, Kandakurti PK, Hazari A. Physical rehabilitation program for cardiorespiratory health and quality of life among breast cancer survivors in UAE: protocol for a randomized control trial. Trials. 2024 Jun 4;25(1):354. doi: 10.1186/s13063-024-08192-9. PMID 38835046